CLINICAL TRIAL: NCT05312788
Title: Effect of Barley Supplemented Wheat Bread on Markers of Cardiovascular and Renal Health: A Randomized Controlled Trial
Brief Title: Effect of Barley Supplemented Wheat Bread on Markers of Cardiovascular and Renal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Bibi Hajira, Assistant Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMU/IBMS/IRBE/2022/9302
Record Dates: First submitted 2022-02-28; First posted 2022-04-06 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Kidney Diseases
Keywords: TBARs; TAC; pCS; Barley; Beta-glucan; E-selectin; NO
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole wheat bread (Placebo Comparator): Whole wheat bread will be used as control bread.
  Interventions: Other: Effect of Barley Supplemented Wheat Bread on markers of Cardiovascular and Renal Health
- Barley supplemented wheat bread (Experimental): Barley supplemented wheat bread (50% substitution) will be used as experimental bread.
  Interventions: Other: Effect of Barley Supplemented Wheat Bread on markers of Cardiovascular and Renal Health

INTERVENTIONS:
Other: Effect of Barley Supplemented Wheat Bread on markers of Cardiovascular and Renal Health — Intervention will involve intake of 50% barley substituted wheat bread.

SUMMARY:
The disruption of colonic microbiota has been linked to a number of diseases, mainly cardiovascular and kidney diseases. One possible means to improve the microbiota is to increase dietary fiber intake as the intake of dietary fiber shifts the fermentation from proteolytic saccharolytic fermentation.

Beta-glucans are soluble dietary fibers mainly found in oats and barley. Results from previous studies suggest that the consumption of barley reduces the risk of cardiovascular and kidney diseases. Therefore, this study will explore the effect of barley beta-glucans on markers of Cardiovascular and Renal health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals of age 18 years or older
* BMI ranged between 18.5 and 24.9

Exclusion Criteria:

* Celiac disease, Cancer, Diabetes , cardiovascular diseases
* Gastro intestinal tract disease
* Pregnant women
* Use of pre-, pro- or antibiotics 15 days before the enrollment into the study
* Food allergy to food used in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Serum Thiobarbituric acid reactive substances (TBARs) from baseline to 4 weeks | Baseline and after 4 weeks
Change in Serum Total antioxidant capacity (TAC) from baseline to 4 weeks | Baseline and after 4 weeks
Change in Serum Nitric oxide from baseline to 4 weeks | Baseline and after 4 weeks
change in Serum E-selectin from baseline to 4 weeks | Baseline and after 4 weeks
Change in Serum P-cresyl sulfate from baseline to 4 weeks | Baseline and after 4 weeks
Change in Serum Indoxyl sulfate from baseline to 4 weeks | Baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Medical University, Peshawar, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosola C, De Angelis M, Rocchetti MT, Montemurno E, Maranzano V, Dalfino G, Manno C, Zito A, Gesualdo M, Ciccone MM, Gobbetti M, Gesualdo L. Beta-Glucans Supplementation Associates with Reduction in P-Cresyl Sulfate Levels and Improved Endothelial Vascular Reactivity in Healthy Individuals. PLoS One. 2017 Jan 20;12(1):e0169635. doi: 10.1371/journal.pone.0169635. eCollection 2017. PMID 28107445
- [Background] Sirich TL, Plummer NS, Gardner CD, Hostetter TH, Meyer TW. Effect of increasing dietary fiber on plasma levels of colon-derived solutes in hemodialysis patients. Clin J Am Soc Nephrol. 2014 Sep 5;9(9):1603-10. doi: 10.2215/CJN.00490114. Epub 2014 Aug 21. PMID 25147155
- [Background] Bacchetti T, Tullii D, Masciangelo S, Gesuita R, Skrami E, Bruge F, Silvestri S, Orlando P, Tiano L, Ferretti G. Effect of a barley-vegetable soup on plasma carotenoids and biomarkers of cardiovascular disease. J Clin Biochem Nutr. 2015 Jul;57(1):66-73. doi: 10.3164/jcbn.15-11. Epub 2015 Jun 5. PMID 26236103
- [Background] Gaesser GA, Rodriguez J, Patrie JT, Whisner CM, Angadi SS. Effects of Glycemic Index and Cereal Fiber on Postprandial Endothelial Function, Glycemia, and Insulinemia in Healthy Adults. Nutrients. 2019 Oct 6;11(10):2387. doi: 10.3390/nu11102387. PMID 31590437